CLINICAL TRIAL: NCT01205594
Title: IRB-HSR# 14296 The Use of the Intrathoracic Pressure Regulator (ITPR) to Improve Systemic Blood Pressure in Patient Undergoing CABG Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Edward C. Nemergut MD, University of Virginia Anesthesiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14296
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: CABG surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITPR device (Experimental): the ITPR will be inserted in the anesthesia circuit and activated to provide -10 mmHg ETP.
  Interventions: Device: ITPR

INTERVENTIONS:
Device: ITPR — the ITPR will be inserted in the anesthesia circuit and activated to provide -10 mmHg ETP.

SUMMARY:
Briefly, after the induction of anesthesia and the placement of TEE, hemodynamic variables (pulmonary and systemic blood pressure, central and pulmonary venous pressure, cardiac output, calculated SVR, etc.) will be collected. In addition, left ventricular performance (including estimates of LVEDV, LVESV, EF, FAC, etc.) will be assessed using TEE. Once these baseline data are recorded, the ITPR will be inserted in the anesthesia circuit and activated to provide -9 mmHg ETP. After the ITPR has been active for at least two minutes, the same hemodynamic and TEE data obtained above will be gathered. After the data is recorded, the ITPR will be disconnected and no further interventions will be made. In addition to the hemodynamic and echocardiographic data described above, an arterial blood gas will be obtained from the pre-existing radial artery catheter during the on- and off- states.

Finally, the TEE examination will be recorded on videotape or DVD. A second echocardiographer, blinded to patient and ITPR status will review each echocardiogram and assess left ventricular performance. In addition to the data derived at the time of testing, the second echocardiographer will assess, if possible, changes in EF using Simpson's method of disks is used to calculate the LV volume.

This is a proof of concept/feasibility study designed to test the primary hypothesis that use of the ITPR will result in increased systemic blood pressure and cardiac output in patients undergoing CABG surgery. The effect of the ITPR on other secondary indicators of cardiac performance will also be examined. These include but are not limited to left ventricular end diastolic volume (LVEDV), ejection fraction (EF), left ventricular end systolic volume (LVESV), and fractional area change (FAC) as assessed by echocardiography, pulmonary artery pressure, and calculated systemic vascular resistance (SVR).

DETAILED DESCRIPTION:
The ITPR is an FDA-approved device intended to increase circulation and blood pressure in hypovolemic and cardiogenic shock. The device is inserted within a standard respiratory circuit between the patient and the ventilator. It functions by decreasing intrathoracic pressure during the expiratory phase to subatmospheric levels after each positive pressure ventilation. The decrease in intrathoracic pressure creates a vacuum within the thorax relative to the rest of the body thereby enhancing blood return to the heart and consequently increasing cardiac output and blood pressure. Activation of the device is also accompanied by a decrease in SVR. The end result is a device that simultaneously improves cardiac output by increasing LVEDP/LVEDV and decreasing SVR while increasing coronary perfusion pressure by increasing blood pressure and decreasing LVESP/LVESV.1-8

ELIGIBILITY:
Inclusion Criteria:

* 1. patients presenting for elective CABG with planned intraoperative TEE 2. age 18 years of age and older 3. informed consent has been obtained

Exclusion Criteria:

* 1. Patients with planned valve surgery (valve or CABG + valve) 2. patients with a contraindication to transesophageal echocardiography (TEE); including patients with extensive esophageal or gastric disease. Relative contraindications include esophageal varices, Barrett's esophagus, Zenker's diverticulum, and postradiation therapy of the esophageal area.

  3. patients requiring IABP or VAD pre-operatively 4. emergent CABG 5. pneumothorax 6. hemothorax 7. uncontrolled bleeding 8. uncontrolled hypertension defined as SBP > 180 mmHg at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
hemodynamic variables | baseline & 2 minutes post device activation
  hemodynamic variables (pulmonary and systemic blood pressure, central and pulmonary venous pressure, cardiac output, calculated SVR) will be collected at baseline & 2 minutes post device activation

SECONDARY OUTCOMES:
left ventricular performance | baseline &2 minutes after activation of the device
  left ventricular performance (including estimates of LVEDV, LVESV, EF, FAC, etc.) will be assessed using TEE.

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Nemergut, MD, Principal Investigator — University of Virginia Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Lurie KG, Zielinski TM, McKnite SH, Idris AH, Yannopoulos D, Raedler CM, Sigurdsson G, Benditt DG, Voelckel WG. Treatment of hypotension in pigs with an inspiratory impedance threshold device: a feasibility study. Crit Care Med. 2004 Jul;32(7):1555-62. doi: 10.1097/01.ccm.0000131207.29081.a2. PMID 15241102
- [Background] Lurie KG, Zielinski T, McKnite S, Aufderheide T, Voelckel W. Use of an inspiratory impedance valve improves neurologically intact survival in a porcine model of ventricular fibrillation. Circulation. 2002 Jan 1;105(1):124-9. doi: 10.1161/hc0102.101391. PMID 11772887
- [Background] Lurie KG, Voelckel WG, Zielinski T, McKnite S, Lindstrom P, Peterson C, Wenzel V, Lindner KH, Samniah N, Benditt D. Improving standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve in a porcine model of cardiac arrest. Anesth Analg. 2001 Sep;93(3):649-55. doi: 10.1097/00000539-200109000-00024. PMID 11524335
- [Background] Lurie KG, Mulligan KA, McKnite S, Detloff B, Lindstrom P, Lindner KH. Optimizing standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve. Chest. 1998 Apr;113(4):1084-90. doi: 10.1378/chest.113.4.1084. PMID 9554651
- [Background] Yannopoulos D, McKnite S, Metzger A, Lurie KG. Intrathoracic pressure regulation improves 24-hour survival in a porcine model of hypovolemic shock. Anesth Analg. 2007 Jan;104(1):157-62. doi: 10.1213/01.ane.0000249047.80184.5a. PMID 17179262
- [Background] Yannopoulos D, McKnite SH, Metzger A, Lurie KG. Intrathoracic pressure regulation for intracranial pressure management in normovolemic and hypovolemic pigs. Crit Care Med. 2006 Dec;34(12 Suppl):S495-500. doi: 10.1097/01.CCM.0000246082.10422.7E. PMID 17114984
- [Background] Yannopoulos D, Metzger A, McKnite S, Nadkarni V, Aufderheide TP, Idris A, Dries D, Benditt DG, Lurie KG. Intrathoracic pressure regulation improves vital organ perfusion pressures in normovolemic and hypovolemic pigs. Resuscitation. 2006 Sep;70(3):445-53. doi: 10.1016/j.resuscitation.2006.02.005. Epub 2006 Aug 9. PMID 16901611
- [Background] Yannopoulos D, Nadkarni VM, McKnite SH, Rao A, Kruger K, Metzger A, Benditt DG, Lurie KG. Intrathoracic pressure regulator during continuous-chest-compression advanced cardiac resuscitation improves vital organ perfusion pressures in a porcine model of cardiac arrest. Circulation. 2005 Aug 9;112(6):803-11. doi: 10.1161/CIRCULATIONAHA.105.541508. Epub 2005 Aug 1. PMID 16061732